CLINICAL TRIAL: NCT05021211
Title: Whole Egg Intake and Choline Concentration in the Aging Brain
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Egg Nutrition Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00146588
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
Keywords: Choline; Egg Consumption; Alzheimer Disease; Cognitive Impairment; Dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Low Egg Consumers: Participants who consume fewer than 1 whole egg per week
- Moderate Egg Consumers: Participants who consume 5-9 whole eggs per week
- High Egg Consumers: Participants who consumes great than or equal to 14 whole eggs per week

SUMMARY:
By doing this study, researchers hope to learn to see if there is relationship between whole egg consumption and brain choline status. Additionally, researchers also plan to see if there is a relationship between brain choline status and cognition.

DETAILED DESCRIPTION:
Participants will come to the research center for 2 different visits. Visit 1 will include anthropometric measurements, surveys, and a cognitive test. Approximately 7-10 days after visit 1, participants will come back to the research center for visit 2. At visit 2, participants will return surveys and a MRI scan will be performed to measure brain choline status. Potential participants need to be located within the Kansas City metro area.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60 - 85 years of age
* Good general health with no concomitant diseases
* Cognitively normal as defined as Mini-mental state examination (MMSE) score ≥ 25
* BMI range: 20 - 40 kg/m2

Exclusion Criteria:

* Presence of central neurological disease (e.g., brain tumor, stroke, epilepsy, motor neuron disease, multiple sclerosis, Alzheimer's, Parkinson's)
* Prior major head trauma with loss of consciousness
* Presence of active unstable and life-threatening illness (e.g., cancer)
* Presence of major psychiatric disorder within the past 3 years including depression, anxiety, and alcohol (over 3 drinks per day or total of 18 per week) or drug abuse (DSM-IV criteria; Geriatric Depression Score > 6)
* Presence of diabetes mellitus or use of anti-diabetic agents
* Use of psychoactive and investigational medications
* Use of hormone replacement therapy
* Tobacco smokers
* Subjects with MRI contraindications

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the greater Kansas City. Recruitment for this research opportunity by email, community flyers, and through the social media platform, Nextdoor. Researchers will also use recruitment databases including the Recruitment and Eligibility Database hosted by the KU Alzheimer's Disease Center (P30 AG035982) and the Pioneers Participant Registry hosted by KU Medical Center and the University of Kansas Hospital. Both of these registries consist of highly characterized, community-dwelling individuals that have given prior consent to be directly contacted for research opportunities.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Association Between Whole Egg Intake and Cerebral Choline | Baseline
  The investigators will recruit a variety of whole egg consumers. Egg consumption will be validated with a 7-day food record 1 week before the MRI. Cerebral choline levels are measured by magnetic resonance spectroscopy (MRS)
Association Between Cerebral Choline and Cognition | Baseline
  The investigators will test the association between cerebral choline as measured by MRS and cognition. Cognition will be measured by the NIH ToolBox cognitive battery.

CONTACTS AND LOCATIONS:
Overall Officials: Debra K. Sullivan, PhD, RD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States